CLINICAL TRIAL: NCT01711021
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover, Laboratory Classroom Study to Evaluate the Safety and Efficacy of d-Amphetamine Transdermal Drug Delivery System (d-ATS) Compared to Placebo in Children and Adolescents With ADHD
Brief Title: Study to Evaluate Safety & Efficacy of d-Amphetamine Transdermal System vs Placebo in Children & Adolescents With ADHD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Noven Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Noven Therapeutics (Industry)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: N25-006
Record Dates: First submitted 2012-10-15; First posted 2012-10-22 (Estimated); Results first posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Dextroamphetamine; Amphetamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- d-Amphetamine Transdermal patch (Active Comparator): The study was conducted in 2 parts: a 5-week, open-label, step-wise Dose Optimization Period and a 2-week, randomized, cross-over Double-Blind Treatment Period.
  Subjects who reached the optimal dose by end of dose optimization treatment period were randomized to receive double-blind treatment.
  Participants first received study patches everyday for one week, then subjects were crossed-over to receive the placebo treatment.
  d-Amphetamine Transdermal System: Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied.
  Interventions: Drug: d-Amphetamine Transdermal Patch
- Placebo patch (Placebo Comparator): The study was conducted in 2 parts: a 5-week, open-label, step-wise Dose Optimization Period and a 2-week, randomized, cross-over Double-Blind Treatment Period.
  Subjects who reached the optimal dose by end of dose optimization treatment period were randomized to receive double-blind treatment.
  Participants first received placebo patches everyday for one week, then subjects were crossed-over to receive the study treatment.
  Placebo patch: Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied.
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: d-Amphetamine Transdermal Patch — The study was conducted in 2 parts: a 5 week, open-label, step-wise Dose Optimization Period and a 2-week, randomized, cross-over Double-Blind Treatment Period.
  Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied.
  Other Names: d-Amphetamine; Amphetamine
  Arms: d-Amphetamine Transdermal patch
Drug: Placebo patch — The study was conducted in 2 parts: a 5 week, open-label, step-wise Dose Optimization Period and a 2-week, randomized, cross-over Double-Blind Treatment Period.
  Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied.
  Other Names: Placebo; Sham treatment
  Arms: Placebo patch

SUMMARY:
This study will evaluate safety and efficacy of d-Amphetamine Transdermal System for the treatment of Attention Deficit Hyperactivity Disorder in children and adolescents.

DETAILED DESCRIPTION:
The study will consist of a four-week screening period, a 3-day wash-out period (if applicable), a five-week open-label, step-wise dose optimization period and two-week double blind randomized crossover treatment period with weekly classroom assessments and a safety follow-up by telephone 7 - 10 days after last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Male or female
2. Age: Between 6 and 17 years of age (inclusive)
3. Race: All eligible
4. Females of child-bearing potential must have agreed to practice a clinically accepted method of contraception during the study and for at least 1 month prior to study dosing and 1 month following completion of the study. Acceptable contraceptive methods included abstinence, oral contraception, surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), intrauterine device, diaphragm in addition to spermicidal foam and condom on male partner, or systemic contraception (e.g., Norplant System)
5. Must have met Diagnostic and Statistical Manual of Mental Disorders, 4th edition - Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD combined, hyperactive/impulsive subtype, or predominately inattentive subtype
6. The Screening and Baseline visit ADHD-RS-IV total score must have been ≥90% of the general population of children by age and gender
7. Able to wear a patch for 9 hours (for children and, if applicable, for adolescents, parent or caregiver must be present to apply and remove the patches and maintain the used and unused patches in a secure, controlled area of the home)
8. Functioning at an age-appropriate level intellectually as determined by an intelligence quotient (IQ) of ≥80 on the Wechsler Abbreviated Scale of Intelligence II™ (WASI II™) vocabulary and matrix reasoning components
9. Must have been able to complete PERMP assessment
10. Must have provided parental consent (signed ICF) and obtained written/verbal assent from the subject
11. Subject and parent(s)/ caregiver must have been willing and able to comply with all the protocol requirements and parent(s) or caregiver must be able to provide transportation for the subject to and from the analog classroom sessions

Exclusion Criteria:

1. Blood pressure outside the 95th percentile for age and gender
2. Pulse of <50 (age 6 - 17), or >120 (age 6 - 12), or >125 (age 13 - 17)
3. Known non-responder to amphetamine treatment
4. Documented allergy, intolerance, or hypersensitivity to amphetamine
5. Currently taking an ADHD medication that is providing symptom control with no residual impairment at home or school and has acceptable tolerability and adherence
6. Recent history (within the past 6 months) of suspected substance abuse or dependence disorder (including nicotine)
7. History of seizures during the last 2 years (excluding infantile febrile seizures), a tic disorder (exclusive of transient tic disorder), a current diagnosis, and/or a family history of Tourette's Disorder. Mild medication-induced tics were not exclusionary
8. Any psychiatric disorder that could interfere with study participation or the safety of the subject or other participants, such as conduct disorder (CD) or oppositional defiant disorder (ODD) with a history of prominent aggressive outbursts. Children meeting CD or ODD but without prominent aggression will be allowed to enroll at the discretion of the Investigator
9. Autism or Asperger's Disorder
10. Family history (first degree relatives) of sudden cardiac death
11. Current controlled (requiring medication) or uncontrolled comorbid psychiatric conditions such as post-traumatic stress disorder, psychosis, bipolar illness, severe obsessive compulsive disorder, severe depressive or severe anxiety disorder, was considered a suicide risk, had recent (last 6 months) suicidal ideation, or any lifetime self-harm event
12. History of abnormal thyroid function
13. Has a body mass index (BMI) for age greater than 95th percentile per Centers for Disease Control BMI (for gender-specific charts)
14. Known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug
15. Any skin abnormality present at the potential application site (i.e., infection, rash, atrophy, excessive fragility or dryness, any cut or abrasion, or tattoo)
16. History of hypersensitivity, allergy to topical medication, preparation, or adhesive dressings
17. Concurrent chronic or significant acute illnesses (such as severe allergic rhinitis or an infectious process requiring antibiotics, unless expected to resolve or has resolved by Day 0) disability or any unstable medical condition that in the Investigator's opinion would lead to difficulty complying with the protocol requirements
18. Used any investigational drug within 30 days of the Screening visit
19. History of physical, sexual, or emotional abuse in the last year
20. Medical history of hepatitis A/B/C or HIV
21. Positive urine drug screen for drugs of abuse

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Waxmonsky, MD, Principal Investigator — Not Affiliated
Locations (3):
- United States (3):
  - University of California - Irvine, Irvine, California
  - Florida International University Center for Children and Families, Miami, Florida
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada

REFERENCES:
- [Derived] Cutler AJ, Suzuki K, Starling B, Balakrishnan K, Komaroff M, Meeves S, Castelli M, Childress A. d-Amphetamine Transdermal System in Treatment of Children and Adolescents with Attention-Deficit/Hyperactivity Disorder: Secondary Endpoint Results and Post Hoc Effect Size Analyses from a Pivotal Trial. J Child Adolesc Psychopharmacol. 2023 Jun;33(5):176-182. doi: 10.1089/cap.2023.0005. PMID 37339441
- [Derived] Cutler AJ, Suzuki K, Starling B, Balakrishnan K, Komaroff M, Castelli M, Meeves S, Childress AC. Efficacy and Safety of Dextroamphetamine Transdermal System for the Treatment of Attention-Deficit/Hyperactivity Disorder in Children and Adolescents: Results from a Pivotal Phase 2 Study. J Child Adolesc Psychopharmacol. 2022 Mar;32(2):89-97. doi: 10.1089/cap.2021.0107. Epub 2022 Jan 11. PMID 35020462

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of 2 study periods. Period 1 is a 5-week open-label Dose Optimization Study with only one arm, Period 2 is a randomized, cross-over, double-blind treatment study (2 weeks).
  A total of 110 subjects were enrolled into the Dose Optimization Treatment (Period 1). 4 subjects did not complete the Dose Optimization Period. 106 subjects were randomized into the Double-Blind Treatment Period (Period 2).
Groups:
- d-Amphetamine Transdermal Patch: The study consisted of 2 study periods. Period 1 is a 5-week open-label Dose Optimization Study with only one arm, Period 2 is a randomized, cross-over, double-blind treatment study (2 weeks). A total of 110 subjects were enrolled into the Dose Optimization Treatment (Period 1). 4 subjects did not complete the Dose Optimization Period. 106 subjects were randomized into the Double-Blind Treatment Period (Period 2).
  Arm Titles are defined for Period 2 (Open-Label Dose Optimization Treatment). For Period 1 study, there is only 1 arm. All participants started with the lowest dose of d-Amphetamine Transdermal System. Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied. Patients return for a visit every week to evaluate whether to increase the dose next week for 5 weeks until an optimized dose was identified. For Period 2 study, participants first received study patches everyday for one week, then subjects were crossed-over to receive the placebo treatment.
- Placebo Patch: Period 1 is open-label, Dose Optimization Treatment Period and has only one treatment arm. No placebo patch were used.
  Placebo Patch was used in Double-Blind Treatment Period, which has 2 arms.
Period: Open-Label Dose Optimization Period
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Started | 110 | 0 (No placebo arm for Period 1 Open-Label Dose Optimization Period.)
Completed | 106 | 0 (No placebo arm for Period 1 Open-Label Dose Optimization Period.)
Not Completed | 4 | 0
Period: Double-blind Cross-Over Treatment Period
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Started | 53 (The 106 subjects who completed Period 1 study (1 arm) were assigned to 2 arms in Period 2 study. Therefore, 53 subjects were assigned to the d-Amphetamine Transdermal Patch, then Placebo arm, another 53 subjects were assigned to the Placebo, then d-Amphetamine Transdermal Patch arm.) | 53 (The 106 subjects who completed Period 1 study (1 arm) were assigned to 2 arms in Period 2 study. Therefore, 53 subjects were assigned to the d-Amphetamine Transdermal Patch, then Placebo arm, another 53 subjects were assigned to the Placebo, then d-Amphetamine Transdermal Patch arm.)
Completed | 46 | 46
Not Completed | 7 | 7

BASELINE CHARACTERISTICS:
Population: A total of 110 subjects entered the Dose Optimization Period. The optimized dose achieved by a subject during this period was then utilized in the Double-Blind Treatment Period of the study. The Demographic and Baseline Characteristics are presented as one arm for all subjects enrolled.
Groups:
- Baseline Characteristics for All Subjects Enrolled: Baseline Characteristics are presented for all subjects that were enrolled (n=110).
Arm/Group | Baseline Characteristics for All Subjects Enrolled
Number analyzed (Participants) | 110
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 110
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.5 (3.09)
Age, Customized [Median (Full Range); unit: years]
  Median Age | 10 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 40
  Not Hispanic or Latino | 70
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 84
  More than one race | 7
  Unknown or Not Reported | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 18.68 (3.369)

OUTCOME MEASURES:

1. Primary Outcome: Mean Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Total Score During the Double-Blind Treatment Period
Description: The SKAMP total score comprises all 13 items. The SKAMP was designed for independent observers to rate 13 items representing 2 factors of classroom behavior: attention (SKAMP-A) and deportment (SKAMP-D), as well as quality of work. Items are specific to place (classroom setting) & time (during a typical classroom period), & the scale is used to assess multiple ratings taken within a day. The SKAMP-D subscale evaluates deportment, including interacting with other children, interacting with adults, remaining quiet according to classroom rules, & staying seated according to classroom rules. The SKAMP-A subscale is a measure of attention & evaluates getting started on assignments, sticking with tasks, attending to an activity, and making activity transitions. The SKAMP quality of work subscale includes 3 items: completing assigned work, performing work accurately, and being careful and neat while writing or drawing. Scores range from 0-78 with higher scores indicating worse impairment.
Time Frame: Mean SKAMP Total Score of SKAMP Total Scores from 9 different time points including (1, 2, 3, 4.5, 6, 7, 9, 10, 12 hours post-dose)
Population: Full Analysis Set: included all consented and randomized subjects who took at least 1 dose of study of medication
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- d-Amphetamine Transdermal Patch: Subjects who reached the optimal dose by end of dose optimization treatment period were randomized to receive double-blind treatment.
  Participants first received study patches everyday for one week, then subjects were crossed-over to receive the placebo treatment.
  d-Amphetamine Transdermal System: Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied.
- Placebo Patch: Subjects who reached the optimal dose by end of dose optimization treatment period were randomized to receive double-blind treatment.
  Participants first received placebo patches everyday for one week, then subjects were crossed-over to receive the study treatment.
  Placebo patch: Patches will be worn for 9 hours every day. After 9 hours the patch will be removed. Every day a new patch will be applied.
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 100 | 101
score on a scale | 12.81 (.32) | 18.67 (.322)
Statistical Analysis 1: Comparison: d-Amphetamine Transdermal Patch vs Placebo Patch; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mixed model repeated measure (MMRM) analysis for SKAMP total score in Double-Blind period; Least Square (LS) mean difference = -5.87, 95% CI 2-sided [-6.76 to -4.97]

2. Secondary Outcome: Onset of Efficacy Measured by Swanson, Kotkin, Agler, M-Flynn, and Pelham (SKAMP) Total Score
Description: Onset of efficacy defined as the time of the first assessment time showing statistical significance between d-ATS and placebo. The time point for the reported data are SKAMP scores (LS mean) from 2 hours post-dose.
  The SKAMP total score comprises all 13 items. The SKAMP was designed for independent observers to rate 13 items representing 2 factors of classroom behavior: attention (SKAMP-A) and deportment (SKAMP-D), as well as quality of work. Items are specific to place (classroom setting) & time (during a typical classroom period), & the scale is used to assess multiple ratings taken within a day. Scores range from 0-78 with higher scores indicating worse impairment.
Time Frame: Onset of efficacy defined as the time of the first assessment time showing statistical significance between d-ATS and placebo. 2 hours post-dose in Double-Blind Treatment Period
Population: Full Analysis Set: included all consented and randomized subjects who took at least 1 dose of study of medication.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 103 | 101
score on a scale | 12.2 (1.01) | 19.0 (1.02)

3. Secondary Outcome: Duration of Effect for d-Amphetamine and Placebo Treatment
Description: Duration of Effect is the difference between the End of Effect and Onset of Effect in hours, where End of Effect is the first time point after Onset of Effect at which the 50% reduction in SKAMP total score from pre-dose is not observed.
Time Frame: Duration of Effect was from onset (2 hours post-dose) and up to 12 hours post-dose (p<0.001)
Population: Full Analysis Set: included all consented and randomized subjects who took at least 1 dose of study of medication.
Measure: Least Squares Mean (Standard Error); unit: Hours
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 61 | 20
Hours | 2.6 (2.08) | 1.7 (0.96)
Statistical Analysis 1: Comparison: d-Amphetamine Transdermal Patch vs Placebo Patch; Test type: Superiority; p = 0.01, Mixed Models Analysis

4. Secondary Outcome: Permanent Product Measure of Performance (PERMP) Scores Including PREMP-C and PREMP-A From Different Timepoints Post-dose
Description: To assess efficacy of d-ATS compared to placebo as measured by the PERMP-C (number of correct answers) and PERMP-A (number of attempted answers) score. The PERMP is an age-adjusted written math test, of 10 minutes' duration administered at multiple time points. Subjects are given 5 pages of 80 math problems (400 total problems) and are instructed to work at their desks and to complete as many problems as possible in 10 minutes. Performance is measured as the number of problems attempted (PERMP-A) and the number of problems worked correctly (PERMP-C). The scores range from 0-800 with higher scores indicating better performance.
Time Frame: 1,2, 3, 4.5,6,7,9,10 and 12 hours post-dose from double-blind treatment period
Population: Full Analysis Set: included all consented and randomized subjects who took at least 1 dose of study of medication
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 106 | 106
score on a scale
  PERMP-C at 1 hour | 124.0 (6.04) | 113.1 (6.07)
  PERMP-C at 2 hours | 139.8 (6.02) | 103.8 (6.07)
  PERMP-C at 3 hours | 141.2 (6.02) | 93.7 (6.07)
  PERMP-C at 4.5 hours | 141.5 (6.02) | 97.9 (6.07)
  PERMP-C at 6 hours | 139.7 (6.02) | 94.3 (6.07)
  PERMP-C at 7 hours | 139.7 (6.02) | 96.2 (6.10)
  PERMP-C at 9 hours | 139.0 (6.07) | 102.9 (6.07)
  PERMP-C at 10 hours | 132.4 (6.07) | 98.9 (6.07)
  PERMP-C at 12 hours | 135.3 (6.07) | 96.4 (6.07)
  PERMP-A at 1 hour | 126.6 (6.07) | 116.3 (6.10)
  PERMP-A at 2 hours | 142.7 (6.04) | 106.3 (6.10)
  PERMP-A at 3 hours | 144.0 (6.04) | 97.4 (6.10)
  PERMP-A at 4.5 hours | 144.0 (6.04) | 100.9 (6.10)
  PERMP-A at 6 hours | 142.0 (6.04) | 96.8 (6.10)
  PERMP-A at 7 hours | 142.3 (6.04) | 98.9 (6.13)
  PERMP-A at 9 hours | 141.7 (6.10) | 106.8 (6.10)
  PERMP-A at 10 hours | 134.7 (6.10) | 102.1 (6.10)
  PERMP-A at 12 hours | 137.4 (6.10) | 100.1 (6.10)

5. Secondary Outcome: Change in the Clinician-rated Scale of ADHD Symptoms Based on DSM-IV-TR Criteria (ADHD-RS-IV).
Description: The ADHD-RS-IV is based on the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria to assess efficacy of d-ATS compared to placebo. The ADHD-RS-IV scale was developed to measure the behaviors of children with ADHD, and it consists of 18 items designed to reflect current symptomatology of ADHD based on DSM-IV criteria. Each item is scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0 to 54.
  Note: Week 6 is the first week of the double-blind treatment period, week 7 is the second week of the double-blind treatment period.
Time Frame: Averaged from week 6 and week 7 results during the Double-Blind Cross-Over treatment period.
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 104 | 106
score on a scale | -23.4 (1.02) | -10.3 (1.02)

6. Secondary Outcome: Conners Parent Rating Scale Revised Short Form (CPRS-R:S) Total Scores From Week 6 and Week 7
Description: The CPRS-R:S evaluates problem behaviors as reported by the parent or alternative caregivers. The CPRS-R:S total score comprises 27 items and covers a subset of the subscales and items on the long parent form. The score ranges from 0-81 calculated from summed subscales scores. Higher score is considered a worse outcome for ADHD patients.
  Note: Week 6 is the first week of the double-blind treatment period, week 7 is the second week of the double-blind treatment period.
Time Frame: Combined analysis by treatment groups from week 6 and week 7 (averaged)
Population: Full Analysis Set Double-Blind period Week 6 and Week 7
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 100 | 100
score on a scale | 23.5 (1.75) | 39.5 (1.75)

7. Secondary Outcome: Number of Responders Evaluated by Clinical Global Impression (CGI-I) Scale by Treatments From the Double-blind Treatment Period
Description: The CGI scale permits a global evaluation of the subject's improvement over time. During the Dose Optimization Period and the Double-Blind Treatment Period, the investigator assessed the subject's improvement relative to symptoms prior to dosing, using the CGI-I Scale.
  For CGI-I scale, the responders are defined as subjects achieving a score of
  1. Very much improved or
  2. Much improved or
     The non-responders are defined as subjects achieving a score of
  3. Minimally improved on the clinician-rated CGI global improvement item or
  4. No change or
  5. Minimally worse or
  6. Much worse or
  7. Very much worse
  Then the number of responders are calculated by treatment arms. Note: Week 6 is the first week of the double-blind treatment period, week 7 is the second week of the double-blind treatment period.
Time Frame: the double-blind treatment period
Population: Responder includes the categories "Very Much Improved" and "Much Improved"; "Non-Responder" includes all other categories, with the exception of "not assessed" which has been considered missing data.
  Note: the Full Analysis Set is 106 (N)
Measure: Count of Participants; unit: Participants
Arm/Group | d-Amphetamine Transdermal Patch | Placebo Patch
Number analyzed (Participants) | 106 | 106
Participants | 89 | 25

ADVERSE EVENTS:
Time Frame: From beginning of Dose-Optimization Phase (5-week) through double blind treatment phase (2-week), up to 7 weeks total.
Groups:
- All d-ATS Treatment During the Dose-Optimization Phase: This includes subjects that started the one arm Dose-Optimization Study in Period 1 and continued into Double-Blind, Cross-Over, Placebo-Controlled Treatment study in Period 2. The adverse events are reported for adverse events including all d-ATS doses during Dose-Optimization Study Phase (Period 1).
- d-ATS Patch Treated Arm During the Double Blind Phase: This includes subjects that started the one arm Dose-Optimization Study in Period 1 and continued into Double-Blind, Cross-Over, Placebo-Controlled Treatment study in Period 2. The adverse events are reported from subjects who received d-ATS patch treatment during the double blind phase.
- Placebo Treated Arm During the Double Blind Phase: This includes subjects that started the one arm Dose-Optimization Study in Period 1 and continued into Double-Blind, Cross-Over, Placebo-Controlled Treatment study in Period 2. The adverse events are reported from subjects who received placebo patch treatment.
Arm/Group | All d-ATS Treatment During the Dose-Optimization Phase | d-ATS Patch Treated Arm During the Double Blind Phase | Placebo Treated Arm During the Double Blind Phase
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/106 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/110 | 0/106 | 0/106
Other Adverse Events (participants affected / at risk) | 108/110 | 44/106 | 32/106
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All d-ATS Treatment During the Dose-Optimization Phase (N=110) | d-ATS Patch Treated Arm During the Double Blind Phase (N=106) | Placebo Treated Arm During the Double Blind Phase (N=106)
Decreased appetite (Metabolism and nutrition disorders) | 64 | 13 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 9 | 4 | 5
Insomnia (Psychiatric disorders) | 29 | 6 | 5
Affect lability (Psychiatric disorders) | 14 | 3 | 0
Initial insomnia (Psychiatric disorders) | 10 | 1 | 0
Irritability (General disorders) | 21 | 2 | 1
Application site pain (General disorders) | 12 | 0 | 0
Fatigue (General disorders) | 10 | 1 | 1
Application site pruritis (General disorders) | 9 | 1 | 1
Pyrexia (General disorders) | 7 | 1 | 1
Headache (Nervous system disorders) | 32 | 6 | 4
Dizziness (Nervous system disorders) | 6 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 13 | 1 | 2
Nasopharyngitis (Infections and infestations) | 11 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 2 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 0 | 3
Abdominal upper pain (Gastrointestinal disorders) | 16 | 3 | 1
Nausea (Gastrointestinal disorders) | 13 | 3 | 1
Vomiting (Gastrointestinal disorders) | 8 | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 7 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2013-05-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT01711021/Prot_000.pdf
  • Statistical Analysis Plan (2013-06-26): https://cdn.clinicaltrials.gov/large-docs/21/NCT01711021/SAP_001.pdf